CLINICAL TRIAL: NCT07399314
Title: Evaluating the Effectiveness of a School-based Stepped Care Treatment Model for Adolescent Depression in Pakistan
Acronym: SMART-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Institute of Human Development (Other)
Collaborators: National Ministry of Health Services, Regulations and Coordination (Unknown); Institute of Psychiatry, Benazir Bhutto Hospital, Rawalpindi (Unknown); Shifa Tameer-e-Millat University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GIHD/Trials/2025/03; ISRCTN11220474 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2026-01-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Depression Anxiety Disorder; Psychological Distress; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: In this sequential multiple assignment cluster randomized controlled trial, randomization will occur in two stages. First, school clusters (N=40), stratified by sex, will be randomized to intervention or control arms in a 1:1 allocation ratio. Schools in the intervention arm will receive the universal socioemotional life skills intervention from non-specialists in classroom settings. It aims at improving socioemotional life skills and providing basic psychological support to adolescents in classroom settings. Adolescents in the control arm will receive Treatment as Usual (TAU). At 3-months from the baseline, a second randomisation will occur at the individual level based on gender and PHQ-9 scores. In both arms, adolescents scoring ≥5 on PHQ-9 will be re-randomised to continue initial treatment (universal or TAU) or a step-up CBT-based guided self-help app.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the interventions, it is not possible to blind adolescents, caregivers, facilitators, supervisors, data managers, or the trial manager. However, assessors, the trial statistician, and investigators will remain blinded. To maintain masking, intervention and assessment teams will operate from separate offices with no interaction. Participants will be instructed not to share their treatment allocation during follow-ups. Masking of fidelity will be assessed by asking assessors to guess participant allocation at the end of each follow-up assessment timepoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Stage Intervention - Universal Intervention for Intervention & TAU for Control Arms (Experimental): The first-stage intervention involves a universal intervention delivered in the intervention arm, while the control arm receives treatment-as-usual (TAU). In the intervention arm, all adolescents aged 13-15 years receive a structured, school-based program delivered by non-specialists. It is grounded in developmental, behavioural, social, and cognitive theories and aims to provide basic psychological support to adolescents, build their socioemotional life skills, and strengthen collaboration between parents and schools, including referral pathways for those requiring specialist care. Using a structured manual, storybooks, and lesson plans, non-specialists deliver interactive sessions in class.
  Mental health services are not available in public schools in Pakistan, so no structured programs will be delivered to adolescents in schools in the control group (TAU).
  Interventions: Behavioral: Universal Intervention & CBT-based Guided Self-Help Application
- Second Stage Intervention - CBT-based self-help app (Experimental): The second-stage intervention in both arms is a CBT-based self-help app. At 3 months from baseline, adolescents scoring ≥5 on PHQ-9 in both arms are individually re-randomised to continue initial treatments (universal intervention/TAU) or receive a step-up, CBT-based guided self-help app. The app, accessible via tablet/mobile, is based on empirically supported strategies.
  Interventions: Behavioral: Universal Intervention & CBT-based Guided Self-Help Application

INTERVENTIONS:
Behavioral: Universal Intervention & CBT-based Guided Self-Help Application — The first-stage intervention is universal intervention in the intervention arm and TAU in the control arm. In the intervention arm, adolescents receive universal intervention from non-specialists, while in the control arm, they receive TAU. Universal intervention, based on developmental, behavioral, social, and cognitive theories, aims to provide basic psychological support to adolescents, build their socioemotional life skills, and strengthen collaboration between parents and schools, including referral pathways for those requiring specialist care. The second-stage intervention is a CBT-based self-help app. At 3-months, adolescents scoring ≥5 on the PHQ-9 in both arms (indicating the presence of depressive symptoms) are individually re-randomized to continue their initial treatment (universal or TAU) or receive a step-up, CBT-based guided self-help app.

SUMMARY:
This study aims to test the effectiveness of a stepped-care model to reduce depressive symptoms in adolescents in school settings in Pakistan. The study will examine whether the universal intervention, delivered by non-specialists, can reduce depressive symptoms in adolescents after 3 months. For adolescents who do not improve with universal intervention, the study will assess whether a Cognitive Behavioural Therapy (CBT)-based guided self-help app can provide additional support as a second-step intervention. Six hundred adolescents aged 13-15 from 40 schools in Rawalpindi, Pakistan, will take part. The study will determine which interventions work best and for which students to reduce depressive symptoms in school settings in Pakistan.

DETAILED DESCRIPTION:
Introduction:

Depression and anxiety symptoms among adolescents can have long-term negative effects on academic, social, and emotional development if not identified and treated early. School-based interventions, both universal and indicated, are recommended to address these symptoms. However, the optimal timing, dosage, and sequencing of such interventions remain unclear, particularly in low-resource settings. The SMART-STEP study in Pakistan aims to address this gap by evaluating two evidence-informed interventions within a stepped-care model: the universal intervention, delivered by trained non-specialists to provide early support to adolescents in schools, and a Cognitive Behavioural Therapy (CBT)-based guided self-help application, designed for adolescents with persistent symptoms. Both interventions are endorsed by the WHO and UNICEF as part of the Helping Adolescent Thrive Toolkit. This study seeks to answer the question, "What works, for whom, under what conditions, and why, for reducing depressive symptoms in adolescents?"

Methods and Analysis:

The investigators will conduct a clustered Sequential Multiple Assignment Randomized Controlled Trial (SMART) to evaluate the effectiveness of these interventions, determine optimal timing and dosage, and identify which students benefit most from which intervention.

Study Setting and Participants: Forty eligible public schools in Rawalpindi, Pakistan, stratified by gender, will be included. Following ethical approvals, adolescents aged 13-15 years will be screened for psychological distress using the Paediatric Symptoms Checklist (PSC). Adolescents scoring above the threshold (≥28 on PSC) will be eligible for the trial. 600 adolescents will be recruited.

Stage 1 Randomisation: Schools and participants will be randomized in a 1:1 allocation ratio into intervention and control arms. The universal socioemotional life skills intervention will be delivered by non-specialists to adolescents in classroom settings.

Stage 2 Randomization: Adolescents who are non-responders at 3 months, defined as PHQ-9 scores ≥ 5, will be individually re-randomised to one of two options:

Continue with the initial intervention or augment with the CBT-based guided self-help app Outcomes: The primary outcome is reduction in depressive symptoms at 9-month from baseline. Secondary outcomes include changes in symptoms of anxiety, psychosocial distress, functioning, and perceived psychological well-being.

Ethics and Dissemination:

Ethics approval has been obtained from the Institutional Review Board of the Global Institute of Human Development, Islamabad, Pakistan. Written informed consent will be obtained from parents or primary caregivers, and assent will be obtained from adolescents. Study findings will be disseminated through peer-reviewed publications, conferences, and community forums.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 13-15 years, currently enrolled in participating schools
2. Provide assent for participation
3. Parental/guardian consent provided
4. Screen positive for psychosocial distress on the youth-reported Pediatric Symptom Checklist (PSC), defined as a total score ≥ 28

Exclusion Criteria:

1. Adolescents who require immediate in-patient (medical and/or psychiatric) care
2. Adolescents with acute protection risks as assessed by a researcher applying the definitions in the WHO mhGAP intervention guide.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2025-11-13 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) for adolescents | Enrollment, 3-months, 6-months and 9-months from baseline
  Depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9) for adolescents, a 9-item instrument rated on a 4-point Likert scale. The total score ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms (worse outcome) over the past 2 weeks. The PHQ-9 has been previously adapted and validated in Pakistan and has demonstrated high internal consistency (Cronbach's α = 0.83).

SECONDARY OUTCOMES:
Paediatric Symptoms Checklist (PSC) | Enrollment, 3-months, 6-months and 9-months from baseline
  The PSC is a 35-item screening scale comprising three subscales: internalizing, externalizing, and attention problems. Items are rated on a 3-point scale, with total scores ranging from 0 to 70. Higher scores indicate greater psychosocial difficulties (worse outcome). The Urdu version of the PSC has been adapted and validated in Pakistan and has demonstrated good reliability and validity.
Revised Children's Anxiety and Depression Scale (RCADS) | Enrollment, 6-months and 9-months from baseline
  This is a 25-item instrument rated on a 4-point Likert scale, with a total transformed score ranging from 0 to 100, used to measure levels of anxiety and low mood. The instrument comprises two subscales (anxiety and depression). Higher scores indicate greater symptom severity (worse outcome). The measure has been adapted and used successfully in Pakistan.
DSM-5 Level 1 Cross-Cutting Symptom Measure | Enrollment, 6-months and 9-months from baseline
  The DSM-5 Level 1 Cross-Cutting Symptom Measure is a self-rated screening instrument that assesses mental health domains relevant across psychiatric diagnoses. It is used to identify additional areas of inquiry that may have a significant impact on the child's treatment and prognosis. Items are rated on a 5-point Likert scale, with higher scores indicating greater symptom severity (worse outcome) over the past 2 weeks.
Checklist of Somatic Symptoms of Distress | Enrollment, 6-months and 9-months from baseline
  The Checklist of Somatic Symptoms of Distress is a 10-item instrument rated on a 3-point Likert scale, with total scores ranging from 0 to 20, used to assess somatic symptoms of distress. Higher scores indicate greater somatic symptom severity (worse outcome). The measure has been previously adapted and used in Pakistan.
Experience of Bullying | Enrollment, 6-months and 9-months from baseline
  Experience of bullying in the past 30 days will be measured using a contextualised version of the Bullying Victimization Questionnaire. The total score ranges from 0 to 12, with higher scores indicating greater levels of peer victimisation (worse outcome).
School Climate | Enrollment, 6-months and 9-months from baseline
  Change in school climate, including students' relationships with teachers, sense of belonging with the school and peers, commitment to school tasks, and participation in school activities, will be measured using an adapted version of the Beyond Blue School Climate Questionnaire (BBSCQ). The questionnaire consists of 28 items, each rated on a 4-point Likert scale, with total scores ranging from 0 to 84. Higher scores indicate a more favourable perception of the school climate (better outcome). The measure will be administered to both adolescents and their caregivers.
Annual Academic Performance and Classroom Attendance | From enrollment to the end of treatment at 9-months]
  Academic performance and classroom attendance will be assessed using official school records, which have been previously used by the investigators in Pakistan. Annual academic performance will be recorded as percentage scores (0-100), with higher scores indicating better academic performance (better outcome). Classroom attendance will be recorded as the percentage of days attended during the academic year (0-100%), with higher percentages indicating better attendance (better outcome).
Short Warwick Edinburgh Mental Wellbeing Scale (SWEMWS) | Enrollment, 6-months and 9-months from baseline
  The Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) is a 7-item self-report measure assessing mental wellbeing, focusing on positive functioning of thoughts and feelings over the past two weeks. Items are rated on a 5-point Likert scale ranging from "none of the time" to "all of the time." Total scores range from 7 to 35, calculated by summing item responses. Higher scores indicate better mental wellbeing (better outcome).
Caregivers' Wellbeing | Enrollment, 6-months and 9-months from baseline
  The Self-Reporting Questionnaire (SRQ) will be used to assess psychological distress, represented by subscales of physical symptoms and emotional symptoms. Items are scored 0 or 1, where a score of 1 indicates the presence of a symptom of psychological distress. Total scores range from 0 to 20, with higher scores indicating greater psychological distress (worse outcome).
Alabama Parenting Questionnaire (APQ) | Enrollment, 6-months and 9-months from baseline
  Parenting practices will be assessed using the Positive Involvement subscale of the Alabama Parenting Questionnaire (APQ). This subscale assesses the extent to which parents engage positively with their children, including friendly communication, involvement in planning and conducting activities, awareness of children's free-time activities, playing games together, helping with homework, interest in day-to-day plans, and knowledge of children's friends. Items are rated on a Likert scale, with higher scores indicating greater positive parental involvement (better outcome).
PSYCHLOPS (Child's psychosocial well-being and functioning) | Enrollment, 6-months and 9-months from baseline
  Child insight into problems and wellbeing will be measured using the self-administered PSYCHLOPS-Kids. The measure assesses three domains: problems, functioning, and wellbeing. PSYCHLOPS-Kids has three versions (pre-therapy, during-therapy, and post-therapy). In this study, the pre-therapy and post-therapy versions will be used as part of the assessment. Domain and total scores are calculated by summing item responses, with higher scores indicating greater problems and poorer wellbeing (worse outcome).
Children's Global Assessment Scale (CGAS) | Enrollment, 6-months and 9-months from baseline
  Global functioning will be assessed using a brief clinician-rated measure that rates adolescents on a scale from 1 to 100, categorised into ten functioning bands. Scores range from 1-10 (indicating severe impairment) to 91-100 (indicating superior functioning). Higher scores indicate better global functioning (better outcome).
The Social Problem-Solving Inventory - Revised Short Form | Enrollment, 6-months and 9-months from baseline
  This is a 25-item instrument rated on a 5-point Likert scale (0-4), used to assess social problem-solving skills, including positive problem orientation, negative problem orientation, rational problem solving, impulsivity-carelessness style, and avoidance style. Total scores are calculated by summing item responses (possible range 0-100). Higher scores indicate better social problem-solving skills (better outcome).
Perceived Emotional/Personal Support Scale | Enrollment, 6-months and 9-months from baseline
  Perceived emotional support will be assessed using a measure rated on a 4-point Likert scale, with scores ranging from 1 to 4, to assess the level of emotional support perceived by the child across three relationship categories: family members, non-family adults, and friends. Higher scores indicate higher levels of perceived emotional support (better outcome).
Client Service Receipt Inventory (CSRI) | Enrollment, and 9-months from baseline
  Health service utilisation will be assessed using a structured measure to collect information on outpatient and inpatient healthcare services used by adolescents over a period of up to 9 months, including contacts with all types of healthcare providers. Higher values indicate greater health service utilisation.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Usman Hamdani, PhD MBBS, Principal Investigator — Global Institute of Human Development
Locations (1):
- Global Institute of Human Development, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The availability of individual participant data (IPD) has not been determined at this time.

REFERENCES:
- [Background] Hamdani SU, Huma ZE, Tamizuddin-Nizami A, Baneen UU, Suleman N, Javed H, Malik A, Wang D, Mazhar S, Khan SA, Minhas FA, Rahman A. Feasibility and acceptability of a multicomponent, group psychological intervention for adolescents with psychosocial distress in public schools of Pakistan: a feasibility cluster randomized controlled trial (cRCT). Child Adolesc Psychiatry Ment Health. 2022 Jun 21;16(1):47. doi: 10.1186/s13034-022-00480-z. PMID 35729589
- [Background] Hamdani SU, Huma ZE, Malik A, Tamizuddin-Nizami A, Javed H, Minhas FA, Jordans MJD, Sijbrandij M, Suleman N, Baneen UU, Bryant RA, van Ommeren M, Rahman A, Wang D. Effectiveness of a group psychological intervention to reduce psychosocial distress in adolescents in Pakistan: a single-blind, cluster randomised controlled trial. Lancet Child Adolesc Health. 2024 Aug;8(8):559-570. doi: 10.1016/S2352-4642(24)00101-9. PMID 39025557
- [Background] Hamdani, S., Huma, Z.E., Javed, H., Warraitch, A., Rahman, A., Nizami, A., & Minhas, F. (2021). Prevalence of psychosocial distress in school going adolescents in rural Pakistan: Findings from a cross-sectional epidemiological survey. BJPsych Open, 7(S1), S56-S57. doi:10.1192/bjo.2021.196
- [Background] Naveed S, Waqas A, Memon AR, Jabeen M, Sheikh MH. Cross-cultural validation of the Urdu translation of the Patient Health Questionnaire for Adolescents among children and adolescents at a Pakistani school. Public Health. 2019 Mar;168:59-66. doi: 10.1016/j.puhe.2018.11.022. Epub 2019 Jan 25. PMID 30685600
- [Background] Spence SH. Structure of anxiety symptoms among children: a confirmatory factor-analytic study. J Abnorm Psychol. 1997 May;106(2):280-97. doi: 10.1037//0021-843x.106.2.280. PMID 9131848
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] D'Zurilla, T. J., Nezu, A. M., & Maydeu-Olivares, A. (1999). Manualfor the Social Problem-Solving Inventory-Revised. North Towanda, NY: Multi-Health Systems
- [Background] Clarke DE, Kuhl EA. DSM-5 cross-cutting symptom measures: a step towards the future of psychiatric care? World Psychiatry. 2014 Oct;13(3):314-6. doi: 10.1002/wps.20154. No abstract available. PMID 25273306
- [Background] Jellinek MS, Murphy JM, Robinson J, Feins A, Lamb S, Fenton T. Pediatric Symptom Checklist: screening school-age children for psychosocial dysfunction. J Pediatr. 1988 Feb;112(2):201-9. doi: 10.1016/s0022-3476(88)80056-8. PMID 3339501
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117